CLINICAL TRIAL: NCT06292884
Title: Establishing Novel Functional Biomarkers for Creatine Deficiency Syndromes
Brief Title: Optical Imaging as a Tool for Monitoring Brain Function in Creatine Deficiency Syndromes
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Other Study IDs: IMAGINER CREATINE
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Creatine Deficiency, X-linked; Creatine Deficiency Syndrome Due to Gamt Deficiency
MeSH Terms: conditions — Creatine deficiency, X-linked; Guanidinoacetate methyltransferase deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CTD affected individuals: Individuals with genetic diagnosis of CTD.
- GAMT-D affected individuals: Individuals with genetic diagnosis of GAMT-D.
- Neurotypical controls: Healthy volunteers without known health or medical issues.

SUMMARY:
The objective of this project is to explore the potential of functional near-infrared spectroscopy (fNIRS) as innovative functional biomarker for clinical trial readiness in Creatine Deficiency Syndromes (CDS), a group of rare neurodevelopmental disorders. Among these disorders, effective treatments are lacking for two. The limited availability of objective and quantitative biomarkers to monitor brain function poses challenges to advancing therapeutic research. With gene therapy trials on the horizon, the need for precise measurement to evaluate treatment efficacy is pressing. This project seeks to address this gap by assessing the prognostic reliability of both resting and task-evoked fNIRS. Arousal of participants will be also assessed through the measure of spontaneous heart rate (HR) fluctuations. The primary objectives of this pilot study are: 1. to determine the feasibility of fNIRS in individuals with CDS; 2. to collect pilot data on individuals with CDS to determine the patterns of cerebral oxygen consumption as measured by fNIRS; 3. to compare cerebral oxygen consumption changes at rest and from visual/auditory tasks in affected individuals versus age-appropriate healthy volunteers. The secondary objectives of this study are: 1. to correlate cerebral oxygen consumption changes from visual/auditory task in affected individuals to other measures of disease state (e.g., neuropsychological assessment, disease- specific severity rating scales); 2. to examine test-retest reliability of our fNIRS measures in both affected individuals and healthy controls.

DETAILED DESCRIPTION:
This is a non-profit study of a cohort of patients with Creatine Deficiency Syndromes genetically determined as CTD, GAMT-D and age-matched healthy controls. The design of the study is observational, case-control. An imaging session using fNIRS (NIRSport2, NIRx Technologies) will be conducted during the visits scheduled for the individual participants. Participants will be assessed for optimal placement of the fNIRS probe on the head through measurement of the fiducial points on the scalp. With the NIRx NIRSPort2 system, the near-infrared sources and detectors are situated in a fabric cap resembling a swim cap that is applied like a hat and secured in place by a velcro chin strap. Once the probe is placed, fNIRS will be measured during a passive viewing/listening task administered on a computer. The montage consists of 8 red light-sources operating at 760 nm and 850 nm, and 7 detectors which can be easily placed into a textile EEG cap (EASYCAP, Herrsching, Germany, size according to head circumference). The systems that are utilized have been selected to be very child-friendly systems, involving no cleaning or abrasion of the scalp preparation and rapid application. Application procedures have been designed to minimize any discomfort to the participant. In parallel, ECG will be collected using the polygraphic input box that integrates the ECG with the fNIRS. ECG records the electrical activity generated by the heart and can be used to derive both the heart rate and the pattern of electrical activity as it moves through the heart. To measure ECG, two electrodes will be applied to the skin over the lower left ribcage and the upper right collar bone after the skin has been cleansed and prepared with either abrasive paper or preparation gel. In total, these measurements should take 30-40 minutes to complete (including application of the NIRS cap). Alongside fNIRS, neuropsychological assessments of affected individuals patients will be conducted. The following outcome measures will be collected assessing: i) cognitive performance (Leiter International Performance Scale, 3rd edition, PPVT-5, simple reasoning tasks on tablets and Vineland Adaptive Behaviour Scale); ii) behavioural disorder (BASC-3 and ABC-2 scales); iii) autistic-like features (SRS-2 and PPD-MRS). The cognitive tasks were chosen to be adapted to the cognitive deficit of affected individuals. A task on tablets with minimal verbal instruction will allow to assess reasoning abilities in severe to moderate ID patients that could not perform classical Wechsler scale (IQ test). Healthy controls will be asked to return 8-12 weeks post their initial visit to undergo repeat fNIRS testing for the purposes of examining test-retest reliability of the fNIRS measurement. If their schedule allows, affected individuals will also undergo repeat fNIRS testing. fNIRS is safe, non-invasive and generally well tolerated. The information obtained from this study will help identify outcome measures for drug testing in future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

CDS participants:

* Age criteria: Between ages 2 years to 50 years old, inclusive at time of enrollment
* Diagnosed with either CTD or GAMT-D with a previously identified pathogenic or likely pathogenic variant in the SLC6A8 or GAMT gene.
* Must also meet the diagnostic criteria for CTD/GAMT-D.
* May be female or male

Typically developing participants:

* Age criteria: Between ages 2 years to 50 years old, inclusive at time of enrollment
* Age- and sex-matched to the CDS participants
* No underlying genetic diagnosis or past/chronic medical condition associated with increased risk for autism spectrum disorder (ASD) and/or ID
* Typical neurodevelopment for age (no established diagnosis or clinical suspicion for ASD or ID)

Exclusion Criteria:

For CDS and Typically developing participants:

* Unwilling or unable to comply with study procedures and assessments
* Contraindications to fNIRS, such as uncooperative or destructive behaviors preventing lead placement or capture by fNIRS equipment
* Traumatic loss of consciousness in the last year
* Has taken an investigational drug as part of another research study, within 30 days prior to study enrollment
* If participant is judged by the PI or Sub-I to be inappropriate for the study for any reason

For Typically developing participants:

* Known or suspected cognitive impairment
* Known history of MRI abnormality
* Current use of psychotropic medications

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Creatine Deficiency Syndromes (CDS) are a family of three rare metabolic disorders (AGAT deficiency, AGAT-D, #602360, GAMT deficiency, GAMT-D, 601240 and Creatine Transporter Deficiency, CTD, #300352) negatively impacting brain development and its function. All CDS share a common, predominantly neurological, clinical presentation, including developmental delay, intellectual disabilities, disturbance of expressive and cognitive speech, psycho-motor impairment, autistic-like behavior, and seizures. Oral Cr supplementation leads to the attenuation of symptoms in AGAT-D patients, while for GAMT-D patients limited improvements can be achieved only at very high dosages. Effective treatments for CTD are completely missing as dietary supplementation with Cr, alone or in combination with its precursors, has very limited success.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Resting-state functional connectivity | 3 years
  The comparison of resting-state fNIRS signal between affected individuals and healthy controls will allow to detect potential alterations of spontaneous brain activity and functional connectivity
Amplitude of sensory-evoked hemodynamic responses | 3 years
  The analysis of the amplitude of sensory-evoked fNIRS signal will allow to assess whether this parameter is able to discriminate between affected individuals and healthy controls. The signal latency will be analysed as well.

SECONDARY OUTCOMES:
Correlation between neurophysiology endpoints and the response on neuropsychological scale. | 3 years
  The correlation analysis will allow to understand whether alterations of functional connectivity and/or sensory-evoked responses can be predictive of the severity of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazziotti R, Scaffei E, Conti E, Marchi V, Rizzi R, Cioni G, Battini R, Baroncelli L. The amplitude of fNIRS hemodynamic response in the visual cortex unmasks autistic traits in typically developing children. Transl Psychiatry. 2022 Feb 8;12(1):53. doi: 10.1038/s41398-022-01820-5. PMID 35136021
- [Background] Scaffei E, Mazziotti R, Conti E, Costanzo V, Calderoni S, Stoccoro A, Carmassi C, Tancredi R, Baroncelli L, Battini R. A Potential Biomarker of Brain Activity in Autism Spectrum Disorders: A Pilot fNIRS Study in Female Preschoolers. Brain Sci. 2023 Jun 14;13(6):951. doi: 10.3390/brainsci13060951. PMID 37371429